CLINICAL TRIAL: NCT02557490
Title: A Randomized Controlled Trial of TACE Hepatic Artery Infusion of Oxaliplatin and Raltitrexed Treatment of Colorectal Cancer With Liver Metastases
Brief Title: Oxaliplatin and Raltitrexed Treatment of Colorectal Cancer With Liver Metastases
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhu Xu (Other)
Responsible Party: Sponsor-Investigator, Zhu Xu, Interventional Therapy Department, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014YJZ16
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-07

CONDITIONS: Colon Cancer Liver Metastasis
Keywords: TACE; hepatic artery infusion; oxaliplatin; raltitrexed
MeSH Terms: interventions — Oxaliplatin; raltitrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxaliplatin by TACE (Experimental): Oxaliplatin for the therapy of Colorectal Cancer With Liver Metastases by TACE.No interventions was raltitrexed for the therapy of Colorectal Cancer With Liver Metastases by TACE.
  Interventions: Drug: oxaliplatin and raltitrexed
- Raltitrexed by TACE (No Intervention): Raltitrexed for the therapy of Colorectal Cancer With Liver Metastases by TACE.

INTERVENTIONS:
Drug: oxaliplatin and raltitrexed — TACE methods: use of epirubicin 20-40mg emulsifier lipiodol embolization target vessel, with gelatin sponge particles or PVA particles or microspheres embolization supplement.
  Hepatic arterial chemotherapy: Bi embolization catheter in the hepatic artery or left hepatic artery branch within the right, chemotherapy, for the experimental group (A group): OXA 130mg / m2 artery 0-4 hours pumped Raltitrexed 3mg/m2 4-5 hours pumped into the arteries; the control group (group B)
  Arms: Oxaliplatin by TACE

SUMMARY:
The purpose of this study was a randomized controlled trial to compare the effect of oxaliplatin and raltitrexed treatment of colorectal cancer with liver metastases by TACE hepatic artery infusion

DETAILED DESCRIPTION:
Colorectal cancer is one of the most common malignancies, with 1 million new cases and half a million deaths each year worldwide. The development of metastases is the main cause of death. Liver metastases are diagnosed in 10-25% of patients at the time of resection of their primary colorectal tumor and, eventually, up to 70% of patients with colorectal cancer develop liver metastases.Oxaliplatin and raltitrexed were used for the treatment of colorectal cancer with liver metastases. We aimed to perform a randomized controlled trial to compare the effect of oxaliplatin and raltitrexed treatment of colorectal cancer with liver metastases by TACE hepatic artery infusion.

ELIGIBILITY:
Inclusion Criteria:

1. With written informed consent
2. Age ranged from 18 to 80 years, both men and women
3. Confirmed by pathology or clinical diagnosis of unresectable colorectal cancer with liver metastases patients(including the primary tumor and liver in patients with brain metastases except outside of metastasis in patients with unresectable)
4. Progress systemic chemotherapy or who can not tolerate chemotherapy, or who refuse chemotherapy
5. Never received TACE treatment
6. (M) RECIST 1.0 criteria measurable liver lesions at several ≥2, each lesion diameter ≥3 cm long and ≤20cm,
7. ECOG PS score of ≤2
8. expected survival time ≥12 weeks
9. The test results before 7 days entered the group must meet the following requirements:

   * Hemoglobin ≥ 90 g / L
   * Absolute neutrophil count (ANC)> 1,500 / mm3
   * Platelet count ≥ 80x109 / L
   * Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <5 times the upper limit of normal (UNL)
   * Total bilirubin <3UNL
   * Serum creatinine <1.5 UNL
   * PT or INR, PPT <1.5 UNL (for patients undergoing warfarin or heparin anticoagulant therapy, if there is no evidence that there is an abnormality of the above parameters, you can enter the group, but must be closely monitored to detect at least once a week until the INR stable)

Exclusion criteria

1. Specific circumstances of patients not suitable for TACE therapy / chemotherapy
2. Hepatic decompensation, or the presence of hepatic encephalopathy
3. Before entering the study with gastrointestinal bleeding within 30 days
4. Presence of brain metastasis
5. Pregnant or lactating women
6. Active bleeding or sepsis
7. History of heart disease:

   * NYHA two or more of congestive heart failure, symptomatic coronary artery disease
   * Need to use β-blockers or digoxin medication other than arrhythmias
8. Despite treatment, still systolic blood pressure> 150 mmHg or diastolic blood pressure> 90 mmHg hypertension
9. Not cure severe trauma, acute or incurable ulcer, or three months fracture
10. The researchers believe their poor compliance
11. Exist once or primary lesion or histologically different tumors and colorectal cancer, except: head and neck carcinoma in situ, cured basal cell carcinoma, superficial bladder cancer (Ta, Tis, T1), and the group 3 years ago, it has been cured of cancer
12. HIV infection or the presence of AIDS-related illness, or severe acute and chronic diseases
13. Drug abuse, or suffering that could interfere with study compliance and other psychological or psychiatric disorders
14. Need drug therapy epilepsy (such as steroids or antiepileptic drugs
15. Chemotherapy contraindications exist
16. Any instability or likely to endanger the patient in this study the safety and compliance of the case

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | three years

SECONDARY OUTCOMES:
overall survival (OS) | three years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Feng AW, Guo JH, Gao S, Kou FX, Liu SX, Liu P, Chen H, Wang XD, Xu HF, Cao G, Zhu X. A randomized phase II trial of hepatic arterial infusion of oxaliplatin plus raltitrexed versus oxaliplatin plus 5-fluorouracil for unresectable colorectal cancer liver metastases. Front Oncol. 2022 Sep 21;12:913017. doi: 10.3389/fonc.2022.913017. eCollection 2022. PMID 36212504